CLINICAL TRIAL: NCT06204458
Title: Evaluation of the Efficacy of Mild Water-filtered Infrared-A Whole-body Hyperthermia to Improve Symptoms and Quality of Life in Patients With Post-COVID Syndrome (HyPoCo)
Brief Title: Mild Water-filtered Infrared-A Whole-body Hyperthermia in Patients With Post-COVID Syndrome (HyPoCo)
Acronym: HyPoCo
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Bavarian State Ministry of Health and Care (Other Government)
Responsible Party: Principal Investigator, Jost Langhorst, Prof. Dr. med., Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23050
Record Dates: First submitted 2024-01-11; First posted 2024-01-12 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-10

CONDITIONS: Post-COVID Syndrome
Keywords: hyperthermia; fatigue; post-COVID syndrome
MeSH Terms: conditions — Hyperthermia; Fatigue

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mild hyperthermia group (Experimental): For the study, the method of passive whole-body hyperthermia is used. The IRATHERM®1000 system (Von Ardenne Institute for Applied Medical Research/Dresden) is used, in which the entire body is heated to a core body temperature above the physiological 37°C under the application of 10L/min oxygen. The aim is to achieve a core body temperature of 38.5°C within the framework of mild whole-body hyperthermia. After this warm-up phase, a temperature plateau phase of about 60 minutes follows, in which an attempt is made to maintain the core body temperature of 38.5°C. In the temperature plateau phase, a slight increase in the body core temperature is usually observed. The total time required for a session is given as 1.5 to 2 hours, but this depends on the individual constitution and daily condition of the patient and can be subject to fluctuations.
  Interventions: Other: mild hyperthermia group
- sham group (Sham Comparator): Within the patient information, privacy policy, etc., there is talk of "gentle hyperthermia" and classic, "mild hyperthermia". This serves to introduce the sham intervention as a control group compared to the patient. Lighting conditions, procedures, instructions and explanations are indistinguishable. Within the application, patients of the sham group will receive a hyperthermia application almost without overheating. In order to achieve this, the patients will be positioned on the IRATHERM®1000 in accordance with the Von Ardenne Institute's regulations. Due to the insulating blanket and the natural device and body heat, the patients of the sham group experience a gentle warmth, which is not the same as regular whole-body hyperthermia and an increase in the body core temperature of about 1.5 °C. In the sham setting, the core body temperature increases by about 0.3 to 0.4 °C within a 55-minute session.
  Interventions: Other: sham group

INTERVENTIONS:
Other: mild hyperthermia group — The hyperthermia treatment is carried out in a cycle of two treatments per week, with at least one day in between, over a period of two weeks, according to the manufacturer's instructions. For better tolerability, the application takes place under administration of 10L/min oxygen. According to the guidelines, the rectal (possibly vaginal) temperature (as body core temperature), heart rate and oxygen saturation (Sp02) are continuously determined during the hyperthermia treatment. During the treatment, continuous supervision by trained personnel is guaranteed, and a doctor is on call.
  Arms: mild hyperthermia group
Other: sham group — Within the application, patients in the Sham group will undergo a hyperthermia application with virtually no overheating. To achieve this, the patients are positioned on the hyperthermia device in the same way as the intervention group. An insulating foil applied beforehand prevents direct irradiation with water-filtered infrared-A radiation. This prevents an increase in temperature. Due to the insulating blanket and the natural heat from the device and body, patients in the Sham group experience a gentle warmth that cannot be compared with regular whole-body hyperthermia and an increase in core body temperature of around 1.5°C. The number of treatments, the lighting conditions and procedures including 10L/min oxygen supply, is equal to the treatments in the intervention group.
  Arms: sham group

SUMMARY:
This study examines the efficacy of mild water-filtered whole-body hyperthermia during outpatient treatment in patients with post-COVID syndrome. The aim is to evaluate whether there can be an improvement in fatigue and quality of life. The duration of the study extends over a treatment period of approximately 2 weeks with two treatment units per week and a follow-up period of 3 months after the outpatient treatment.

DETAILED DESCRIPTION:
A total of about 60 participants over 18 years of age are sought, who will be divided into two groups of equal size after inclusion in the study. All participants will receive the same amount of water-filtered whole-body hyperthermia (WBH) under application of 10 L/min oxygen within the outpatient setting. One group receives the gentle form of WBH, the other group receives the classic, mild WBH, which differ in the intensity of the radiation. Gentle hyperthermia serves as a control group for mild hyperthermia.

All abnormalities are documented by the responsible therapists, doctors and nurses.

Blood parameters are collected before the start, after 2 applications and after the last application during the clinical stay. The aim here is to determine the differential blood count and inflammatory and immune parameters; among other things, autoantibody production is to be examined and monitored during the course of the study. In order to check the possible effectiveness of the treatment, various questionnaire values are also collected. The survey will take place at 3 points in time (at the beginning, after completion of the 4 treatments and 3 months afterwards).

In addition, a diary will be filled out in which patients will provide information on their sleep, personal energy level and pain level as well as their daily step count in order to create an activity profile. All patients receive a paper diary and a pedometer adapted to their individual characteristics in advance. The diary is to be kept from week 0 to week 15.

After completion of the study, qualitative interviews lasting around 30-45 minutes will be conducted with 16-20 participants in weeks 8-10 of the follow-up period. Participants are selected on the basis of socio-demographic and clinical characteristics with the aim of obtaining a sample that is as heterogeneous as possible. The interviews are conducted by telephone.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years
* Confirmed diagnosis of post-COVID syndrome
* Fatigue: at least 51.5 points on the MFI-20 scale.
* Signed declaration of consent

Exclusion Criteria:

* Participation in other clinical studies
* Contraindications for hyperthermia (severe cardiovascular diseases with/above NYHA II, active tumor diseases, acute infections, hyperthyroidism (not adjusted), pregnant and breastfeeding women, epilepsy, high-grade cardiac arrhythmia including atrial fibrillation, multiple sclerosis, major skin lesions, photosensitivity disease, acute exacerbated bronchial asthma/COPD [Gold II to IV])
* Pleuritic chest pain
* Hyperthyroidism
* Poorly controlled diabetes mellitus
* Condition after critical illness due to COVID-19
* Patients with active tumor disease, with pneumological, rheumatic, endocrine or neurological concomitant diseases (including dementia, epilepsy, multiple sclerosis), in particular neurological diseases associated with cognitive or sensory disorders
* Severe liver or kidney diseases (liver cirrhosis, post liver transplant, autoimmune hepatitis, dialysis patients, post kidney transplant, acute kidney failure, autoimmune nephropathy)
* Patients with chronic cannabis use (exception: CBD for myalgia), long-term use of WHO class III opioids (e.g. for myalgia/joint pain), long-term use of immunosuppressive medication (steroids, biologics, MTX, leflunomide, azathioprine)
* Patients with psychiatric disorders (bipolar disorder, psychosis, schizophrenia, personality disorder)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-20 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Multidimensionl Fatigue Inventory (MFI-20) | Week 0
  An inventory including 20 questions about fatigue-symptoms (each from 1 ("Yes, that is true") to 5 ("No, that is not true")) covering 5 dimensions (general fatigue, physical fatigue, reduced motivation, reduced activity, mental fatigue).
Multidimensionl Fatigue Inventory (MFI-20) | Week 3
  An inventory including 20 questions about fatigue-symptoms (each from 1 ("Yes, that is true") to 5 ("No, that is not true")) covering 5 dimensions (general fatigue, physical fatigue, reduced motivation, reduced activity, mental fatigue).

SECONDARY OUTCOMES:
Multidimensionl Fatigue Inventory (MFI-20) | Week 15
  An inventory including 20 questions about fatigue-symptoms (each from 1 ("Yes, that is true") to 5 ("No, that is not true")) covering 5 dimensions (general fatigue, physical fatigue, reduced motivation, reduced activity, mental fatigue).
Brief Pain Inventory (BPI) - Intensity of pain (Numeric Rating Scale, NRS) | Week 0
  An inventory including 15 Items about the intensity of pain (4 items, numeric rating scales from 1 (no pain) to 10 (worst pain imaginable); primary outcome), pain impairment (7 items with NRS from 1-10) and the efficacy of medications/treatments.
Brief Pain Inventory (BPI) - Intensity of pain (Numeric Rating Scale, NRS) | Week 3
  An inventory including 15 Items about the intensity of pain (4 items, numeric rating scales from 1 (no pain) to 10 (worst pain imaginable); primary outcome), pain impairment (7 items with NRS from 1-10) and the efficacy of medications/treatments.
Brief Pain Inventory (BPI) - Intensity of pain (Numeric Rating Scale, NRS) | Week 15
  An inventory including 15 Items about the intensity of pain (4 items, numeric rating scales from 1 (no pain) to 10 (worst pain imaginable); primary outcome), pain impairment (7 items with NRS from 1-10) and the efficacy of medications/treatments.
Pittsburgh Sleep quality index (PSQI) | Week 0
  An inventory including 10 questions (plus subquestions) about the quality of sleep. Most of the questions range from ("Not during the past month" to "thee or more times a week"). The questions can be calculated in seven subscales.
Pittsburgh Sleep quality index (PSQI) | Week 3
  An inventory including 10 questions (plus subquestions) about the quality of sleep. Most of the questions range from ("Not during the past month" to "thee or more times a week"). The questions can be calculated in seven subscales.
Pittsburgh Sleep quality index (PSQI) | Week 15
  An inventory including 10 questions (plus subquestions) about the quality of sleep. Most of the questions range from ("Not during the past month" to "thee or more times a week"). The questions can be calculated in seven subscales.
Generic quality of life | Week 0
  Short Form SF-12 Health Survey Questionnaire; A low total value correlates with a poor quality of life, a higher one with a better one.
Generic quality of life | Week 3
  Short Form SF-12 Health Survey Questionnaire; A low total value correlates with a poor quality of life, a higher one with a better one.
Generic quality of life | Week 15
  Short Form SF-12 Health Survey Questionnaire; A low total value correlates with a poor quality of life, a higher one with a better one.
Quality of life (EQ-5D) | Week 0
  The EQ-5D measures 5 dimensions of quality of life (mobility, self-care, general activities, pain/physical discomfort and anxiety/depression) as well as the general state of health on a VAS from 0-100.
Quality of life (EQ-5D) | Week 3
  The EQ-5D measures 5 dimensions of quality of life (mobility, self-care, general activities, pain/physical discomfort and anxiety/depression) as well as the general state of health on a VAS from 0-100.
Quality of life (EQ-5D) | Week 15
  The EQ-5D measures 5 dimensions of quality of life (mobility, self-care, general activities, pain/physical discomfort and anxiety/depression) as well as the general state of health on a VAS from 0-100.
Anxiety and Depression | Week 0
  Hospital Anxiety and Depression Scale (HADS), 14 items (7 each for depressive symptoms or symptoms of anxiety). The two summated scores of the summated scales HADS-A and HADS-D range between 0 and 21. High scores indicate depressivness and anxiety.
Anxiety and Depression | Week 3
  Hospital Anxiety and Depression Scale (HADS), 14 items (7 each for depressive symptoms or symptoms of anxiety). The two summated scores of the summated scales HADS-A and HADS-D range between 0 and 21. High scores indicate depressivness and anxiety.
Anxiety and Depression | Week 15
  Hospital Anxiety and Depression Scale (HADS), 14 items (7 each for depressive symptoms or symptoms of anxiety). The two summated scores of the summated scales HADS-A and HADS-D range between 0 and 21. High scores indicate depressivness and anxiety.
G-EEE (Generic Rating for Treatment pre-experiences, Treatment Expectations and Treatment effects) | Week 0
  A non validated inventory including 11 items measuring pre-experiences, treatment expectations and treatment effects.
G-EEE (Generic Rating for Treatment pre-experiences, Treatment Expectations and Treatment effects) | Week 3
  A non validated inventory including 11 items measuring pre-experiences, treatment expectations and treatment effects.
G-EEE (Generic Rating for Treatment pre-experiences, Treatment Expectations and Treatment effects) | Week 15
  A non validated inventory including 11 items measuring pre-experiences, treatment expectations and treatment effects.
Perceived Stress (PSS-10) | Week 0
  Perceived stress is determined using the Perceived Stress Scale (PSS). The PSS is an international standard instrument for recording subjective stress levels. The official German 10-item version is used in the study.
Perceived Stress (PSS-10) | Week 3
  Perceived stress is determined using the Perceived Stress Scale (PSS). The PSS is an international standard instrument for recording subjective stress levels. The official German 10-item version is used in the study.
Perceived Stress (PSS-10) | Week 15
  Perceived stress is determined using the Perceived Stress Scale (PSS). The PSS is an international standard instrument for recording subjective stress levels. The official German 10-item version is used in the study.
Canadian consensus criteria (CCC) | Week 0
  This is a questionnaire for the diagnosis of CFS/ME (Carruthers et al. 2003). This definition scheme can be used to clinically confirm the diagnosis of CFS/ME. The list of criteria includes the following symptom complexes: Fatigue, exercise intolerance (PEM), sleep disturbances, pain, neurological or cognitive symptoms, autonomic symptoms, neuroendocrine symptoms and immunological symptoms.
Patient Interview | Week 8-10
  Qualitative telephone interviews with 16-20 patients of the mild whole-body hyperthermia group (Experimental group) to get detailed experiences of the patients (30-45 min).
Adverse events (AE) | Week 1-2
  Description of adverse events during the interventions by therapists.
Patient Diary | Week 1-15
  Documentation of pain progression, energy level, sleep, medication intake, number of steps, adverse events
Pedometer (step count) | Week 1-15
  Individual activity profile

OTHER OUTCOMES:
Blood count | Week 0
  (to measure baseline status)
Blood count | Week 2
  (to measure acute effects)
Blood count | Week 3
  (to measure acute effects)
C-reactive Protein (CRP) | Week 0
  Level of C-reactive protein (CRP) in blood to measure inflammation
C-reactive Protein (CRP) | Week 2
  Level of C-reactive protein (CRP) in blood to measure inflammation
C-reactive Protein (CRP) | Week 3
  Level of C-reactive protein (CRP) in blood to measure inflammation
Blood cell sedimenation rate (BSG) | Week 0
  to measure inflammation
Blood cell sedimenation rate (BSG) | Week 2
  to measure inflammation
Blood cell sedimenation rate (BSG) | Week 3
  to measure inflammation
Cytokine panel | Week 0 - baseline status
  Plasma levels of cytokines (TNF-a, IL-6, IL-8, IL-10, etc.)
Cytokine panel | Week 2 - before 3rd application of hyperthermia
  Plasma levels of cytokines (TNF-a, IL-6, IL-8, IL-10, etc.)
Cytokine panel | Week 3 - after last application of hyperthermia
  Plasma levels of cytokines (TNF-a, IL-6, IL-8, IL-10, etc.)
post-Covid autoantibodies | Week 0 - baseline status
  blood parameter
post-Covid autoantibodies | Week 2 - acute effects
  blood parameter
post-Covid autoantibodies | Week 3 - acute effects
  blood parameter
Post-Covid pathogen reactivation | Week 0 - baseline status
  pathogens EBV, CMV, VZV, Pan-/Corona; analysis by Elispot method
Post-Covid pathogen reactivation | Week 3 - acute effects
  pathogens EBV, CMV, VZV, Pan-/Corona; analysis by Elispot method
Real time deformability cytometry (RT-DC) | Week 0 - baseline status
  Blood cell characterization
Real time deformability cytometry (RT-DC) | Week 3 - acute effects
  Blood cell characterization

CONTACTS AND LOCATIONS:
Overall Officials: Jost Langhorst, Prof. Dr., Principal Investigator — Sozialstiftung Bamberg
Locations (1):
- Sozialstiftung Bamberg, Bamberg, Germany